CLINICAL TRIAL: NCT01646190
Title: Fast-Track Perioperative Care After Elective Colorectal Surgery in Senior Patients. Randomized Controlled Trial
Brief Title: Fast-Track Colorectal Surgery in Senior Patients
Acronym: FT-SS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Sandrine Ostermann, Senior Registrar in Digestive Surgery / MD, PhD, swiss board in surgery (FMH), University Hospital, Geneva
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: NAC 08-060
Record Dates: First submitted 2012-07-18; First posted 2012-07-20 (Estimated); Last update posted 2012-07-23 (Estimated); Status verified 2012-07

CONDITIONS: Colorectal Disorders
Keywords: Fast-track; multimodal perioperative care; enhanced recovery; colorectal surgery; elderly patients; seniors
MeSH Terms: interventions — Fluid Therapy; Preanesthetic Medication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard care (Active Comparator): Preoperative: Fasting state after midnight, no intake of oral carbohydrate load Preanesthetic medication No preoperative utilization of inspirex Intraoperative: Effective perioperative analgesia Routine nasogastric tube and abdominal drainage at surgeon discretion Postoperative: Removal of the nasogastric tube after return of bowel function removal of abdominal drainage at surgeon discretion or if volume <50cc Oral liquids and stepwise oral nutrition (water to others liquids to progressive normal or low-fiber nutrition Switch to oral medication after oral nutrition tolerance Urinary catheter removal when the mobilization is satisfactory Mobilization: non standardized and encouraged stepwise mobilization Discharge criteria discussed at surgeon discretion
  Interventions: Behavioral: Fasting state after midnight; Other: Preanesthetic medication
- FT perioperative care (Experimental): Preoperative carbohydrate load No preanesthetic medication General anesthesia and intravenous analgesia Transoesophageal US-Doppler for individualized i.v fluids therapy POD 0: No Nasogastric tube postoperatively Oral liquids 0.3-0.5L 6h after extubation First mobilization 6h after surgery (2h) Stimulation of inspirex utilization (6-8t/d) POD 1: Free oral liquids; progressive normal or low-fiber diet Switch to oral medication Urinary catheter removal Mobilization: >4 h out of bed (walking, chair) inspirex utilization POD 2: Free oral liquids; normal or low-fiber diet Mobilization: >6 h out of bed (walking, chair), inspirex utilization POD 3: Complete mobilization as preoperatively First evaluation of discharge criteria in the afternoon
  Interventions: Dietary Supplement: Preoperative Carbohydrate load; Procedure: individualized i.v fluids therapy; Behavioral: No Nasogastric tube postoperatively; Behavioral: urinary catheter removal; Behavioral: Oral liquids; Behavioral: Stimulation of inspirex utilization; Behavioral: Mobilization

INTERVENTIONS:
Dietary Supplement: Preoperative Carbohydrate load — oral intake in the evening before surgery and 2-3h before intubation
  Arms: FT perioperative care
Procedure: individualized i.v fluids therapy — by Transoesophageal aortic US-Doppler done intraoperatively
  Arms: FT perioperative care
Behavioral: Fasting state after midnight — No preoperative glucose load
  Arms: Standard care
Behavioral: No Nasogastric tube postoperatively — Withdrawal after complete awakening in operating room
  Arms: FT perioperative care
Behavioral: urinary catheter removal — at POD 1
  Arms: FT perioperative care
Behavioral: Oral liquids — 0.3-0.5L oral liquids at 6h postoperatively on POD 0
  Arms: FT perioperative care
Behavioral: Stimulation of inspirex utilization — using 6-8 times/day to prevent pulmonary atelectasis
  Arms: FT perioperative care
Behavioral: Mobilization — First active mobilization 6h after surgery (2h on chair or 45° sitting in bed), >4h out of bed on POD1, >6h on POD2, complete at POD3
  Arms: FT perioperative care
Other: Preanesthetic medication — Preanesthetic oral medication before surgery
  Arms: Standard care

SUMMARY:
Fast-track (FT) surgery is a multimodal, multidisciplinary-team approach to reduce perioperative surgical stress and injury after colorectal surgery, resulting in lower morbidity and enhanced recovery. As fast-track approach could probably be the most beneficial for senior patients to reduce postoperative morbidity and better preserve independency, only scarce information is available in senior population. Therefore a randomized controlled trial is initiated in our institution compare a senior dedicated fast-track approach to modern standard care after colorectal surgery.

DETAILED DESCRIPTION:
BACKROUND:

The multimodal concept of fast-track (FT) surgery was developed by Kehlet et al. in the 1990s to reduce perioperative surgical stress after colorectal surgery, resulting in lower morbidity & mortality and enhanced recovery.

The main evidence-based FT components include: pain control optimization by epidural or systemic analgesia, short-acting anesthetics, opioids-sparing analgesia, minimally invasive surgery, preoperative carbohydrate administration, normothermia preservation, individualized i.v goal-directed fluids therapy, no bowel preparation, no routine use of drains, nasogastric tube, urinary catheters, early oral nutrition and active ambulation, as well as a dedicated preoperative counseling defining the FT clinical pathway and discharge criteria.

Many cohort studies, randomized controlled trials, meta-analyses and systematic reviews have demonstrated its safety and efficacy for decreasing morbidity, hospital stay, and improving patient satisfaction as compared to standard care (SC).

Only scarce information, mainly based on RetroPro or controlled clinical trials (CCTs), is available on fast-track perioperative care in senior patients (>70 years) as they already represent 15-18% of western population, and over 40% of colorectal surgeries performed at Geneva University Hospital (HUG).

The aim of this randomized controlled trial (RCT) is to compare short-term clinical outcomes of a specifically senior designed fast-track perioperative program versus standard care (SC) after elective colorectal surgery in senior patients.

OBJECTIVES:

30-day postoperative morbidity according to Dindo-Clavien classification of complication is the primary clinical endpoint.

Length of hospital stay (LOS) including readmission, autonomy preservation (through the activities of daily living (ADLs) and instrumental activities of daily living (IADL) scale) and quality of life evaluation are secondary endpoints.

METHOD:

All patients over 70 years requiring elective colorectal surgery will be included in this study after given written informed consent. Exclusion criteria consisted in emergency revisional or liver-associated surgery, and inability to discern/speak French or English. Patients will be 1:1 randomized (institutional table of randomization.

ELIGIBILITY:
Inclusion Criteria:

* senior patients (> or = 70 years at operation)
* elective colorectal surgery

Exclusion Criteria:

* emergency, liver-associated, revisional surgeries
* inability to discern or speak French/English, dementia
* absolute contraindication to systemic analgesia (severe allergic reaction)

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2009-12; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
30-day morbidity according to Dindo-Clavien classification | Postoperative day (POD) 0 to 30
  Dindo-Clavien classification of postoperative complication (Grade I to V), including mortality (grade V)

SECONDARY OUTCOMES:
Length of hospital stay (LOS) | discharge day
  LOS: from operating date to discharge
quality of life (QoL) | POD 0, 30 at 6 and 12 months
  QoL using a validated questionnaire for digestive surgery (SF-12) 0 to 44 points for 7 items
readmission | until POD 30
  readmission in any hospital for any reason during the 30 postoperative days
Level of independance | POD 0, 30, at 6 and 12 months
  using geriatric functional scale: ADLs(0-6), IADLs (0-7)scoring

OTHER OUTCOMES:
Pain evaluation | POD 0 at 6h and 24h, POD 2, POD 3
  Pain score through visual analogue scale (VAS)
Fatigue évaluation | POD 0 at 6h and 24h, POD 2, POD 3
  Fatigue measured through numeric scale:0 (no fatigue) to 3 (severe) fatigue

CONTACTS AND LOCATIONS:
Overall Officials: Sandrine Ostermann, MD, PhD, Principal Investigator — University Hospital, Geneva
Locations (1):
- University Hospital, Geneva, Geneva, Switzerland

REFERENCES:
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Derived] Ostermann S, Morel P, Chale JJ, Bucher P, Konrad B, Meier RPH, Ris F, Schiffer ERC. Randomized Controlled Trial of Enhanced Recovery Program Dedicated to Elderly Patients After Colorectal Surgery. Dis Colon Rectum. 2019 Sep;62(9):1105-1116. doi: 10.1097/DCR.0000000000001442. PMID 31318772
- See also: University Hospital Geneva official website for senior surgery — http://visceral-surgery.ch/visceral/index.php?option=com_content&view=article&id=307&Itemid=179&lang=fr